CLINICAL TRIAL: NCT06495073
Title: Determining the Minimal Clinically Important Difference (MCID) for the TOPICS-SF and PROMIS-10 in Older Patients That Suffered an Ischemic Stroke or Transient Ischemic Attack (TIA), Using an Anchor-based Approach
Brief Title: Determining the MCID for the TOPICS-SF and PROMIS-10 in Older Patients That Suffered an Ischemic Stroke or TIA
Acronym: CONSIDER
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. dr. Nathalie van der Velde, Full Professor Geriatric medicine (internal medicine), Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA), Amsterdam UMC, location AMC
Other Study IDs: 2023.0822
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-10

CONDITIONS: Ischemic Stroke; TIA
Keywords: MCID; PROMIS-10; TOPICS-SF
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PROMIS-10 and TOPICS-SF — There will be no intervention. The participants will be asked to fill in questionnaires at two time points: the first time will be after informed consent when they are at the hospital for diagnostic evaluation of the TIA or ischemic stroke, and the second time will be 4 weeks later, with a window of 2 weeks (allowing a range of 2-6 weeks). The second time point is chosen because the investigators suspect that by then, around 50% will be in the "improved" group. At the first time point, the participants will be asked to fill in the PROMIS-10 and element D and E of the TOPICS-SF - which are the elements used to determine the functional limitations and the psychological wellbeing. At the second time point, the participants will be asked to answer the same questions, as well as three additional anchor questions.

SUMMARY:
Patient-related outcome measures (PROMs) play a crucial role in assessing patient outcomes in healthcare. Two of these PROMs are the The Older Persons and Informal Caregivers Survey Short Form (TOPICS-SF) and Patient-Reported Outcomes Measurement Information System Global Health Short Form (PROMIS-10). The investigators aim to determine the Minimal Clinically Important Difference (MCID) for the TOPICS-SF and PROMIS-10 in older people that suffered an ischemic stroke or Transient Ischemic Attack (TIA), using an anchor-based method.

DETAILED DESCRIPTION:
Patient-related outcome measures (PROMs) play a crucial role in assessing patient outcomes in healthcare. Two of these PROMs are the TOPICS-Short Form (TOPICS-SF) and PROMIS Global Health-10 (PROMIS-10). The TOPICS-SF, a shortened version of the TOPICS MDS, is a 20-item survey used in geriatric medicine to collect data on daily functioning. The PROMIS-10, a 10-question survey, is a global measure of the mental and physical health of stroke survivors.

The Minimal Clinically Important Difference (MCID) for PROMs is used to determine the clinical significance of differences in patients' scores. The MCID is defined as "the smallest difference in score in the domain of interest which patients perceive as beneficial and which would mandate, in the absence of troublesome side effects and excessive cost, a change in the patient's management".

MCID values vary across different populations. Despite the significance of MCID in interpreting PROM results, neither TOPICS-SF nor PROMIS-10 have established MCID values for the population of older adults that suffered a stroke.

One option to determine the MCID for these PROMs is a distribution-based method: this method compares the change in scores on the PROMS to statistical measures of spread of the data like the standard deviation. However, this approach may not always provide clinically relevant differences. A method that provides a more clinically meaningful MCID estimate is the anchor-based method.

With the anchor-based method, a specific question or "anchor" is chosen that is related to the concept being measured by the PROM. This anchor question typically asks participants about their perceived change in health or well-being over a specified period. For example, it might be a question like, "Has your physical health improved since ….?" The response options often include choices like "yes/no" or a range of improvement levels. The PROMs and the anchor questions are administered to the same group of participants, both before and after a specific time period. Based on the responses to the anchor question, participants are categorized into different groups like "improved" and "not improved". The MCID is then calculated using the predictive modeling approach. This technique uses statistical modeling techniques to analyze the relationship between changes in PROM scores and the categories established by the anchor question. The MCID value obtained through this process represents the minimum change in PROM scores that is considered clinically significant from the participant's perspective.

The investigators aim to determine the MCID for the TOPICS-SF and PROMIS-10 in people aged 70 or older that suffered an ischemic stroke or Transient Ischemic Attack (TIA), using an anchor-based method, to determine the clinical significance of differences in participant' scores.

This will be achieved through a prospective cohort study with no intervention. Participants will complete questionnaires at two time points: initially after providing informed consent during their hospital visit for diagnostic evaluation of the TIA or ischemic stroke, and then again four weeks later (with a two-week window, allowing for a range of two to six weeks). At the first time point, participants will complete the PROMIS-10 and elements D and E of the TOPICS-SF, which assess functional limitations and psychological well-being. At the second time point, participants will answer the same questions along with three additional anchor questions. The MCID for the PROMIS-10 and TOPICS-SF will be calculated using prognostic modeling techniques.

ELIGIBILITY:
Inclusion Criteria:

* age = 70 years or older at the time of ischemic stroke or TIA;
* inclusion within a week after diagnosis of ischemic stroke or TIA

Exclusion Criteria:

* not speaking Dutch;
* being unable to answer questions;
* being unable or not willing to give written informed consent.

Ages: 70 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The patient population consists of older (>=70 yrs) patients with a recent acute ischemic stroke or TIA who are admitted to or Amsterdam UMC location AMC or the OLVG West hospital, or visit the outpatient clinic or emergency department of one of these hospitals for diagnostic evaluation. Diagnosis of ischemic stroke or TIA will be left to the discretion of the neurologist.
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
MCID of the PROMIS-10 | 4 weeks
  The Minimal Clinically Important Difference (MCID) of the Patient-Reported Outcomes Measurement Information System Global Health Short Form(PROMIS-10) will be calculated using an achor-based approach. The PROMIS-10 has scores ranging from 10 to 50, where higher scores indicate better health status.
MCID of the TOPICS-SF | 4 weeks
  The Minimal Clinically Important Difference (MCID) of the The Older Persons and Informal Caregivers Survey Short Form (TOPICS-SF) will be calculated using an achor-based approach. Of the TOPICS-SF, the investigators will use the questions regarding physical and psychological wellbeing (section D and E). These sections have combined scores ranging from 0 (worst) to 54 (best).

SECONDARY OUTCOMES:
MCID of the mental health score of the PROMIS-10 | 4 weeks
  Since the Patient-Reported Outcomes Measurement Information System Global Health Short Form(PROMIS-10) provides subscales for mental health (ranging from 4 to 20 points, higher scores indicating better mental health), as well as a global measure of the health related quality of life, the investigators will try to calculate the The Minimal Clinically Important Difference (MCID) for the mental health subscale.
MCID of the physical health score of the PROMIS-10 | 4 weeks
  Since the Patient-Reported Outcomes Measurement Information System Global Health Short Form(PROMIS-10) provides subscales for physical health (ranging from 4 to 20 points, higher scores indicating better physical health), as well as a global measure of the health related quality of life, the investigators will try to calculate the The Minimal Clinically Important Difference (MCID) for the physical health subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Renske van den Berg-Vos, Prof, dr., Principal Investigator — Amsterdam UMC, Academic Medical Center, University of Amsterdam, Amsterdam, The Netherlands; Nathalie van der Velde, Prof, dr, Principal Investigator — Amsterdam UMC, Academic Medical Center, University of Amsterdam, Amsterdam, The Netherlands
Locations (2):
- Netherlands (2):
  - OLVG, locatie West, Amsterdam, North Holland
  - Amsterdam UMC, locatie AMC, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: Yes
The CONSIDER database can be requested by other researchers. These requests will be reviewed according the requirements for sharing CONSIDER data.
Supporting Information: Study Protocol
Time Frame: After data-collection/analysis.
Access Criteria: privacy laws of the Netherlands, including policy of NFU and AmsterdamUMC must be followed:
  * data will be shared anonymously
  * data can only be used to study the research question for which participants signed the ICF
  * data will not be shared for commercial purposes.